CLINICAL TRIAL: NCT03650517
Title: A Prospective Observational Multi-center 4 Cohort Study Comparing Robotic Assisted and Laparoscopic Invasive Right Colectomy and Intracorporeal Anastomosis Versus Extracorporeal Anastomosis
Brief Title: Minimally Invasive Right Colectomy Anastomosis Study
Acronym: MIRCAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Other Study IDs: IDIVAL CI18/27
Record Dates: First submitted 2018-07-16; First posted 2018-08-28 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer; Anastomotic Complication; Colectomy
Keywords: Laparoscopic; Robotic; Right colon tumor; Anastomosis; Intracorporeal; Extracorporeal
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Robotic Surgical Procedures; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Robotic Right Colectomy with ICA: Robot-assisted surgery (RAS), allows many types of complex MIS procedures using robotic systems to aid in surgical procedures providing more precision, flexibility and control than is possible with other MIS techniques.
  Intracorporeal anastomosis: when the anastomosis is performed inside the abdominal cavity with a laparoscopic or robotic technique. A Pfannenstiel incision will be done exclusively for specimen extraction.
  Interventions: Procedure: Intracorporeal Anastomosis; Procedure: Robotic Surgery
- Robotic Right Colectomy with ECA: Robot-assisted surgery (RAS), allows many types of complex MIS procedures using robotic systems to aid in surgical procedures providing more precision, flexibility and control than is possible with other MIS techniques.
  Extracorporeal anastomosis: when the anastomosis is performed by pulling out the bowel through a laparotomy wherever that laparotomy is performed.
  Interventions: Procedure: Extracorporeal Anastomosis; Procedure: Robotic Surgery
- Laparoscopic Right Colectomy with ICA: Laparoscopic surgery, also called minimally invasive surgery (MIS), or keyhole surgery, is a surgical technique in which operations are performed far from their location through small incisions (usually 0.5-1.5 cm) elsewhere in the body.
  Intracorporeal anastomosis: when the anastomosis is performed inside the abdominal cavity with a laparoscopic or robotic technique. A Pfannenstiel incision will be done exclusively for specimen extraction.
  Interventions: Procedure: Intracorporeal Anastomosis; Procedure: Laparoscopic Surgery
- Laparoscopic Right Colectomy with ECA: Laparoscopic surgery, also called minimally invasive surgery (MIS), or keyhole surgery, is a surgical technique in which operations are performed far from their location through small incisions (usually 0.5-1.5 cm) elsewhere in the body.
  Extracorporeal anastomosis: when the anastomosis is performed by pulling out the bowel through a laparotomy wherever that laparotomy is performed.
  Interventions: Procedure: Extracorporeal Anastomosis; Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Extracorporeal Anastomosis — Anastomosis is performed by pulling out the bowel through a laparotomy wherever that laparotomy is performed.
  Groups: Laparoscopic Right Colectomy with ECA; Robotic Right Colectomy with ECA
Procedure: Intracorporeal Anastomosis — Anastomosis is performed inside the abdominal cavity with a laparoscopic or robotic technique
  Groups: Laparoscopic Right Colectomy with ICA; Robotic Right Colectomy with ICA
Procedure: Robotic Surgery — Procedure is performed using robotic instruments
  Groups: Robotic Right Colectomy with ECA; Robotic Right Colectomy with ICA
Procedure: Laparoscopic Surgery — Procedure is performed using standard laparoscopic instruments
  Groups: Laparoscopic Right Colectomy with ECA; Laparoscopic Right Colectomy with ICA

SUMMARY:
Right colectomy (hemicolectomy) involves the removal of the cecum, the ascending colon, the hepatic flexure, the first one-third of the transverse colon, part of the terminal ileum, and the associated regional fat and lymph nodes, and is the accepted treatment for malignant neoplasms of the right colon.

A minimally invasive approach is commonly used for right colectomy, with studies reporting reduced complications, less blood loss, and hospital stay when compared to an open approach.

However, there remains controversy regarding whether robotic assistance is advantageous for this technique and whether an intracorporeal (ICA) or extracorporeal anastomosis (ECA) is best.

MIRCAST is a prospective, observational, international, multi-center, 4-parallel-cohorts study. Sites or surgeons will select a cohort of the study for which they are qualified. Four cohorts will be the subject of study:

1. Robotic Right Colectomy with ICA
2. Robotic Right Colectomy with ECA
3. Laparoscopic Right Colectomy with ICA
4. Laparoscopic Right Colectomy with ECA

All patient assessments will be done according to the sites standard of care. Parameters routinely recorded during right colectomy surgery will be collected prospectively. Enrolled subjects will undergo assessments at the following intervals: pre-operative, operative, discharge, 30 days, 3 months, 1 year and 2 years post-surgery.

DETAILED DESCRIPTION:
MIRCAST study is an observational, prospective, parallel cohorts, international, multi-center to compare robotic assisted and laparoscopic minimally invasive right colectomy, and intracorporeal anastomosis versus extracorporeal anastomosis.

The research is coordinated by Marcos Gómez Ruiz MD PhD from Hospital Universitario Marqués de Valdecilla in Santander, Spain; the sponsorship is performed by Fundacion Instituto de Investigación Marqués de Valdecilla (IDIVAL). The European Society of Coloproctology (ESCP) endorses MIRCAST Study and will run a quality audit/independent monitoring of the study.

The objectives of study are to compare of the peri-operative complications after robotic assisted and laparoscopic minimally invasive right colectomy with intracorporeal anastomosis versus extracorporeal anastomosis.

To Identify potential benefits of robotic assisted procedures for right colon resections.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Right colon tumor with indication for right colectomy (benign or malignant disease)
* Patient has a life expectancy of at least 12 weeks
* Patients with adequate performance status (Eastern Cooperative Oncology Group Scale score of ≤2)
* Patient has signed and dated the Informed consent before patient inclusion in the study

Exclusion Criteria:

* Patient with a comorbid illness or condition that would preclude the use of surgery
* Patients with cT4b tumors
* Patients unwilling to comply with all follow-up study requirements
* Patient undergoing emergency procedures
* Planned colonic surgery along with major concomitant procedures (e.g. liver resections, other intestinal resections)
* Metastatic disease
* Pregnant or suspected pregnancy
* Inflammatory Bowel Disease (Crohn´s Disease or Ulcerative Colitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Right colon tumor with indication for right colectomy
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Surgical wound infection | 30 days
  (CDC definition [Health Protection Agency. Surveillance of Surgical Site Infection in England: October 1997-September 2005. London: Health Protection Agency; 2006): Superficial incisional, affecting the skin and subcutaneous tissue. These infections may be indicated by localised (Celsian) signs such as redness, pain, heat or swelling at the site of the incision or by the drainage of pus.
Clavien Dindo Complication | 30 days
  Complications according to Clavien Dindo Classification.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive
Disease Free Survival (DFS) | 2 years
  Length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.
Local Recurrence rate | 2 years
  Rate of cancer that has recurred at or near the same place as the original (primary) tumor
Distant metastases rate | 2 years
  Rate of Cancer that has spread from the original (primary) tumor to distant organs or distant lymph nodes
Rate of Unplanned Conversions to open surgery | 7 days
  When anything apart of the anastomosis had to be done through the laparotomy. If the anastomosis is not completely performed in an intracorporeal approach, the case is considered also converted
Operative time (min) | 7 days
  Operative time from skin to skin in minutes
Complete mesocolic excision (CME) | 30 days
  Complete Mesocolic Excision is defined as complete resection of the mesocolon with its anatomical envelope. Anatomical report should include any defect on CME specimen (Hohenberger W, Weber K., Matzel K., Papadopoulost T., Merkel S. Standardized surgery for colonic cancer: complete mesocolic excision and central ligation - technical notes and outcome. Colorectal Disease 11, 354-365 2008. doi:10.1111/j.1463-1318.2008.01735.x)
Number of Harvested Lymph Nodes | 30 days
  Number of harvested Lymph nodes according to the definitive pathological report.
R0 Resection | 30 days
  Rate of resection without any affected margins during the surgical procedure.
Length of Stay (LOS, days) | 3 months
  In hospital stay of the patient from the day that they are admitted before surgery to the day that they are fit to leave the hospital after the procedure.
Ventral hernia (assessed 1& 2 years after the right colectomy) | 1 and 2 years after the procedure
  Incidence of ventral hernia 1 year after the procedure and 2 years after the procedure at the laparotomy site.
Quality of Life Questionnaire (QLQ) of the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 | 3 months and 1 year after the procedure
  Quality of Life Questionnaire (QLQ) of the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 Score 3 months and 1 year after the procedure.
Quality of Life Questionnaire (QLQ) of the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-CR29 | 3 months and 1 year after the procedure
  Quality of Life Questionnaire (QLQ) of the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-CR29 Score 3 months and 1 year after the procedure.
C-Reactive Protein value (CRP) days 1 & 3 postoperative | 1 and 3 postoperative days.
  CRP values on postoperative day 1 and 3.

OTHER OUTCOMES:
Procalcitonine (PCT) days 1, 3 & 5 postoperative | 1, 3 and 5 postoperative days
  PCT values on postoperative dates 1, 3 and 5
Time to deambulation | 30 days
  Time until patient gets out of bed and engages in light activity (such as sitting, standing, or walking)
Return to work/activity | 30 days and 3 months
  o Time to start working/activity at patient´s job again
Pain evaluation | Postoperative days 1, 3 and 5
  Visual analogue scale (VAS) scores at postoperative days. Scores will range from 0 to 10 (0 no pain and 10 a pain you would rather prefer to die).

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Gómez Ruiz, MD PhD, Principal Investigator — Hospital Universitario Marqués de Valdecilla, IDIVAL; Galo Peralta, MD, Study Chair — Instituto de Investigación Marqués de Valdecilla
Locations (32):
- County Hospital Požega, Požega, Croatia
- Denmark (2):
  - Hospital of Southern Denmark, Aabenraa
  - Zealand University Hospital, Køge
- Finland (5):
  - Kanta-Hämeen Keskussairaala, Hämeenlinna
  - Kymenlaakso Central Hospital, Kotka
  - Päijät-Häme Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
- France (5):
  - Hôpital Haut-Lévèque- CHU, Bordeaux
  - CHU Estaing, Clermont-Ferrand
  - ICM - Institut Régional du Cancer de Montpellier, Montpellier
  - CHRU de Strasbourg Hôpital Civil, Strasbourg
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
- Medizinische Hochschule Hannover, Hanover, Germany
- Eurokliniki Athinou, Athens, Athina, Greece
- Italy (6):
  - AOU-Careggi, Florence
  - Ospedale La Misericordia, Grosseto
  - IEO - European Institute of Oncology, Milan
  - Policlínico Agostino Gemelli, Roma
  - Humanitas Research Hospital, Rozzano
  - IRCCS Istituto di Candiolo, Torino
- Centro Hospitalar de Leiria, Leiria, Portugal
- Spain (9):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Vall d´hebron, Barcelona, Catalonia
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Complejo hospitalario de Torrecardenas, Almería
  - Hospital de León, León
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de octubre, Madrid
- Portsmouth Hospital NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez Ruiz M, Bianchi PP, Chaudhri S, Gerjy R, Gogenur I, Jayne D, Khan JS, Rautio T, Sanchez-Guillen L, Spinoglio G, Ulrich A, Rouanet P. Minimally invasive right colectomy anastomosis study (MIRCAST): protocol for an observational cohort study of surgical complications using four surgical techniques for anastomosis in patients with a right colon tumor. BMC Surg. 2020 Jul 13;20(1):151. doi: 10.1186/s12893-020-00803-x. PMID 32660467